CLINICAL TRIAL: NCT06872359
Title: Prospective, Multicentric, Open Label Clinical Investigation to Evaluate Performance and Safety of Injectable KIO017 Device Range for Facial Tissue Filling
Brief Title: Evaluation of Performance and Safety of Injectable KIO017 Device Range for Facial Tissue Filling
Acronym: LITCHEE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kiomed Pharma (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-1174-U5
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Dermal Fillers; Cheek Augmentation; Lip Augmentation; Perioral Rhytids; Mid-facial Volume Deficit Related to Aging; Lip Enhancement; Lip Augmentation and Correction of Perioral Rhytids; Volume Deficiency in the Mid-Face; Volume Loss of the Jawline; Jawline Definition; Contouring; Midface Contour Deficiencies; Nasolabial Fold Improvement; Nasolabial Folds Correction; Facial Wrinkles; Facial Rhytides
Keywords: Filler; Carboxymethyl chitosan; Hyaluronic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (KIO017-1) (Experimental): Subject seeking an improvement in at least one of the following indications: chin retrusion, mid-face deficit, jawline ptosis
  Interventions: Device: KIO017-1
- Group 2 (KIO017-2) (Experimental): Subject seeking an improvement in at least one of the following indications: temple volume deficit, moderate to severe nasolabial folds, moderate to severe marionette lines, mid-face deficit
  Interventions: Device: KIO017-2
- Group 3 (KIO017-3) (Experimental): Subject seeking an improvement in lip volume/contour and/or perioral lines.
  Interventions: Device: KIO017-3

INTERVENTIONS:
Device: KIO017-1 — Subcutaneous and/or supraperiostal injections in chin and/or mid-face and/or jawline. One (1) injection session on D0 and one (1) touch-up session on M1. The total volume injected per face and per session will not exceed 8 ml.
  Arms: Group 1 (KIO017-1)
Device: KIO017-2 — Subcutaneous injections in temples and/or nasolabial folds and/or marionette lines and/or mid-face. One (1) injection session on D0 and one (1) touch-up session on M1. The total volume injected per face and per session will not exceed 8 ml.
  Arms: Group 2 (KIO017-2)
Device: KIO017-3 — Injections in or around labial mucosa for lip volume and contour and/or intradermal injections in perioral lines. One (1) injection session on D0 and one (1) touch-up session on M1. The total volume injected per face and per session will not exceed 8 ml.
  Arms: Group 3 (KIO017-3)

SUMMARY:
The goal of this clinical trial is to primarily evaluate the performance of KIO017 in filling/volumizing after injection in different areas in healthy women or men, older than 18 years and seeking an improvement of her/his face aspect with resorbable filler. The main questions it aims to answer are:

If the products are safe

- Acceptable local tolerance, with acceptable clinical signs after injection.

If the clinical performance is as intended compared to baseline

* Evaluation of performance by assessing the improvement of the appearance of the defect to be corrected by using Global Aesthetic Improvement Scale (GAIS)
* Quantification of the improvement using the appropriate scale when available or other appropriates tool (angle for chin, for instance).
* Pain felt during injection and after injection
* Subject satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subject
* Sex: male or female
* Age: more than 18 years
* Subject seeking an improvement of her/his face aspect with resorbable filler

  * The subjects must meet a criterion according to the treatment indication specific scale (Asher Face Volume Loss Scale (FVLS), Bazin Ptosis of the Lower part of the Face Scale (PLFS), temple hollow scale (THS), Wrinkle Severity Rating Scale (WSRS), Bazin Marionette Lines scale (MLS), Bazin Upper Lip Wrinkle Scale (ULWS), Rossi scale)
* Subject having given their free, express, and informed consent
* Subject psychologically able to understand the information related to the study, and to give their written informed consent
* Subject affiliated to a health social security system
* Women of childbearing potential should use a contraceptive method considered effective since at least 12 weeks and throughout the study
* Women of childbearing potential must have a negative urinary pregnancy test on D0

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship
* Subject in a social or sanitary establishment
* Subject participating to another clinical research or being in an exclusion period for a previous study
* In France: subject having received 6000 euros indemnities for participation in clinical research in the 12 previous months, including participation in the present study
* Subject already included in another group of this study
* Subject having received treatment with a laser, ultrasound or radiofrequency treatment, a dermabrasion, a surgery, a chemical peeling or any other procedure based on active dermal response on the face in the 6 previous months
* Subject having received mesotherapy products or botulinum toxin in the same area in the 6 previous months
* Subject having received resorbable filling product (e.g., hyaluronic acid) injections in the same area in the 12 previous months
* Subject having received slowly resorbable filling product (e.g., calcium hydroxyapatite, polycaprolactone, polylactic acid) injections in the same area or resorbable threads in the 24 previous months
* Subject having received injections of permanent products in the face (e.g., acrylate polymers, silicone, polytetrafluoroethylene)
* Subject having received facial or cervico-facial lifting in the 24 previous months
* Subject wearing skin support device (mesh, gold threads, permanent lifting threads) on the face
* Subject with uncontrolled and/or recently recovered (<6 months) depression or psychiatric disorders or any other disorder that may pose a health risk to the subject in the study and/or may have an impact on the study assessments
* Subject with severe, ongoing and uncontrolled diseases such as malignancy or history of malignancy, type I diabetes, liver failure, renal failure, lung/heart disease, neoplasia, malignant blood disease, HIV, or other major disease (e.g., systemic fungal infection)
* Subject with recurrent porphyria, untreated epilepsy, coronary insufficiency, ventricular rhythm disorders, severe hypertension, obstructive cardiomyopathy, hyperthyroidism
* Subject with any skin or systemic disease (acute and/or chronic), in the previous year, likely to interfere with the measured parameters or to put the subject to an undue risk
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency
* Subject with current cutaneous inflammatory or infectious processes (e.g., acne, herpes, mycosis, papilloma, chronic eczema, atopic dermatitis …), abscess, unhealed wound, or a cancerous or precancerous lesion on the face
* Subject with multiple allergies, anaphylactic shock history, evolutive allergic pathologies, history of granulomatous diseases
* Subject with known hypersensitivity to chlorhexidine
* Subject having history of allergy or hypersensitivity to one of the components of the tested device, like hyaluronic acid, lidocaine or other amine-type local anaesthetics. polysaccharides of edible mushrooms
* Subject predisposed to keloids or hypertrophic scarring
* Subject with coagulation and/or homeostasis disorders
* Subject with evidence of lymphatic or venous stasis or serious blood disorders
* Subject with pigmentation disorders
* Subject with history of Streptococcus disease (recurrent sore throats, acute rheumatic fever)
* Subjects with congenital methemoglobinemia or receiving concomitant treatment with methaemoglobin-inducing agents
* For subject injected in the chin: subject with clinically significant malocclusion (severe overbite), having dentures and/or any device covering the palate that would interfere with visual assessment of the chin area
* Subject with tattoos, piercings, facial hairs mole or scar that would interfere with visual assessment on the injected area
* Subject with symptoms consistent with COVID-19 or suffering from ongoing symptoms from previous COVID-19 infection
* Subject under anti-coagulant treatment (such as aspirin, nonsteroidal anti-inflammatory drugs) or treatment liable to interfere with the healing process or hemostasis, within 1 month prior to injection, and one-month post-injection.
* Subject with a treatment that reduces or inhibits hepatic metabolism (cimetidine, beta-blockers, etc..)
* Subject having received a vaccine within 21 days prior to injection or planning to do in the 14 days post-injection
* Subject having received dental care within 6 weeks prior to the study or planning to have dental care within 6 weeks post-injection
* Subject receiving any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject to undue risk
* Subject undergoing a topical (on the face) or systemic treatment:

  1. anti-inflammatory medication and/or antihistamines within 2 weeks prior to injection, and 1 month post-injection
  2. corticosteroids within 1 month prior to injection, and 1-month post-injection
  3. retinoids and/or immunosuppressors within 3 months prior to injection and during the study
* Intensive exposure to sunlight or UV-rays within the previous month and/or planning to do so during the study
* Heavy smoker (subject who reports smoking 10 or more cigarettes per day);
* Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of improvement of KIO017 device range on GAIS (Global Aesthetic Improvement Scale) | The measurement is performed on Month 3 after the injection
  Proportion of indications having an improvement with the overall KIO017 range of devices as assessed by the investigator in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of Safety | Evaluation is performed on the Month 1 after injection.
  Assessment of number and percentage of subjects with Adverse Device Effects (ADEs). ADEs are defined as any adverse event related to the use of the investigational medical device.

SECONDARY OUTCOMES:
Assessment of proportion of indications having an improvement on GAIS (Global Aesthetic Improvement Scale) by the investigator in live | Measurement of improvement after injection on the Month 1, Month 6, Month 9, Month 12, Month 18 and Month 24
  Proportion of indications having an improvement with the overall KIO017 range of devices as assessed by the investigator in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of each product and proportion of indications having an improvement on GAIS (Global Aesthetic Improvement Scale) by the investigator in live | Measurement of improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  For each product, proportion of indications having an improvement with each KIO017 device as assessed by the investigator in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of each indication and proportion of subjects having an improvement on GAIS (Global Aesthetic Improvement Scale) by the investigator in live | Measurement of improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  For each indication, proportion of subjects having an improvement with each KIO017 device as assessed by the investigator in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of proportion of indications having an improvement on GAIS (Global Aesthetic Improvement Scale) by the subject in live | Measurement of improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  Proportion of indications having an improvement with the overall KIO017 range of devices as assessed by the subject in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of each product, proportion of indications having an improvement on GAIS (Global Aesthetic Improvement Scale) by the subject in live | Measurement of improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  For each product, proportion of indications having an improvement with each KIO017 device as assessed by the subject in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of each indication, proportion of subjects having an improvement on GAIS (Global Aesthetic Improvement Scale) by the subject in live | Measurement of improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  For each indication, proportion of subjects having an improvement with each KIO017 device as assessed by the subject in live using the GAIS (in 5 points from "worse" (5) to very much improved" (1))
Assessment of improvement on Bazin Ptosis of the Lower part of the Face Scale (PLFS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on Bazin Ptosis of the Lower part of the Face Scale (PLFS) for the subjects injected in jawline with KIO017-1 (in 6 grades: from grade 0 to grade 5)
Assessment of the improvement via glabella-subnasal-pogonion facial angle | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on glabella-subnasal-pogonion facial angle for the subjects injected in chin with KIO017-1
Assessment of improvement on Ascher Face Volume Loss Scale (FVLS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on Ascher Face Volume Loss Scale (FVLS) for subjects injected in mid-face with KIO017-1 or KIO017-2 (in 5 grades: from grade 1 to grade 5)
Assessment of improvement on Temple Hollow Scale (THS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on a descriptive Temple Hollow Scale (THS) for subjects injected in temples with KIO017-2 (in 5 grade: from grade 0 to grade 4)
Assessment of improvement on Wrinkle Skin Rating Scale (WSRS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on a Wrinkle Skin Rating Scale (WSRS) for subjects injected in nasolabial folds with KIO017-2 (in 5 grades: from from 1 to grade 5)
Assessment of improvement on Bazin Marionette Lines Scale (MLS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24
  Change from baseline and proportion of subjects with improvement based on a Bazin Marionette Lines Scale (MLS) for subjects injected in marionette lines with KIO017-2 (in grade 7: from grade 0 to grade 6)
Assessment of improvement on Rossi scale | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 9, Month 12 (for upper lip and lower lip)
  Change from baseline and proportion of subjects with improvement based on a Rossi scale for subjects injected in lips with KIO017-3 (in grade 5: from grade 1 to grade 5)
Assessment of performance on Bazin Upper Lip Wrinkle Scale (ULWS) | Measurement of change/proportion of subjects with improvement after injection on the Month 1, Month 3, Month 6, Month 9 and Month 12
  Change from baseline and proportion of subjects with improvement based on a Bazin Upper Lip Wrinkle Scale (ULWS) for subjects injected in perioral lines with KIO017-3 (in grade 7: from grade 0 to grade 6)
Assessment of average pain on Visual Analog Scale (VAS) | One hour after the last injection and each day for two days after each injection session
  Assessment of average pain felt by the subjects during each injection session using a 0-100 mm VAS
Assesmment of injector satisfaction via questionnaire | Questionnaire completed immediately after each injection session: Day 0, Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  Description in percentages of injector's satisfaction on the injection and instruction for use quality using a questionnaire (in grade 5: from "very satisfied" to "very dissatisfied")
Assessment of subject satisfaction via questionnaire | On Day 0 before the injection and at each timepoint: Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  Description in percentages of satisfaction of the subjects with the treatment using a subjective evaluation questionnaire
Assessment of local tolerance on Injection Site Reactions (ISRs) scale reported by the subjects | During one month after each injection session on the daily-log: Day 0, Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  Description of the number, maximum severity and duration of ISRs reported by the subjects (in 4 grade: from grade 0 to grade 3)
Assessment of local tolerance on Injection Site Reactions (ISRs) scale evaluated by the investigator | On Day 0 after the injection and after each injection session: on Month 1, Month 3, Month 6, Month 9, Month 12, Month 18 and Month 24
  Description of ISRs evaluated by the investigator (in 4 grade: from grade 0 to grade 3)
Number of AEs (Adverse Effects) and ADEs (Adverse Device Effects) | From the first injection and till the Month 24
  Collection of AEs (Adverse Effects) and ADEs (Adverse Device Effects)

CONTACTS AND LOCATIONS:
Overall Officials: Siham Rharbaoui, Dr, Principal Investigator — Eurofins Dermscan Pharmascan
Locations (3):
- France (2):
  - Eurofins Dermscan Pharmascan, Aix-en-Provence
  - Eurofins Dermscan Pharmascan, Villeurbanne
- Centrum Medyczne "Tu Sie Leczy", Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided